CLINICAL TRIAL: NCT03571048
Title: Pilot Study of Time Restricted Feeding as a Weight Loss Intervention in Overweight and Obese Adults
Brief Title: Pilot Study of Time Restricted Feeding as a Weight Loss Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-0487; R21DK117499-02 (NIH)
Record Dates: First submitted 2018-05-31; First posted 2018-06-27 (Actual); Results first posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced Calorie Diet (RCD) (Active Comparator): Participants in this group will focus on daily calorie restriction as their dietary weight loss strategy.
  Interventions: Behavioral: Reduced Calorie Diet (RCD)
- Time Restricted Feeding (TRF) (Experimental): Participants in this group will focus on time restricted feeding in addition to daily calorie restriction as their dietary weight loss strategy.
  Interventions: Behavioral: Reduced Calorie Diet (RCD); Behavioral: Time Restricted Feeding (TRF)

INTERVENTIONS:
Behavioral: Reduced Calorie Diet (RCD) — Participants will be given an individualized calorie goal. Participants in this group will also receive a 12 week comprehensive group-based behavioral weight loss program and will be instructed in specific strategies to support RCD.
Behavioral: Time Restricted Feeding (TRF) — Participants will be given an individualized calorie goal. Participants in this group will also receive a 12 week comprehensive group-based behavioral weight loss program and will be instructed in specific strategies to support RCD. Participants in this group will also instructed to eat only during a window of 10 hours, starting within 3 hours of waking. They will also be instructed in specific strategies to support TRF including: strategies to deal with hunger outside eating windows, distraction techniques, and choosing a balanced diet/appropriate portions during feeding windows.
  Arms: Time Restricted Feeding (TRF)

SUMMARY:
The circadian timing of Energy Intake (EI) has emerged as a key factor in the regulation of body weight. Studies have suggested that eating later in the evening or at night when the circadian system is promoting sleep adversely influences weight loss. In contrast, restricting EI to a short window during waking hours and extending the length of the overnight fast (i.e., time restricted feeding, TRF) may be a practical and useful weight loss strategy. The overall objective of this proposal is to provide a foundation to inform the design of a future large-scale trial to evaluate the efficacy of TRF in generating weight loss. The investigators aims are to: 1) Assess processes critical for the success of a large-scale trial comparing the efficacy of a reduced calorie diet with time restricted feeding (RCD+TRF) versus standard RCD on weight loss; 2) Develop methodology to assess compliance to the RCD+TRF versus standard RCD program and collect preliminary data on whether the programs have differential effects on free-living behaviors (EI, appetite, physical activity, and sedentary behavior); and 3) Measure metabolic responses to RCD+TRF versus standard RCD to determine candidate mechanisms related to weight loss at 12wks and weight maintenance at 6mo post-intervention. The investigators primary hypothesis is that weight loss will be greater in the TRF group compared to the RCD group.

DETAILED DESCRIPTION:
The circadian timing of energy intake (EI) has emerged as a key factor in the regulation of body weight. Studies have suggested that eating meals later in the evening or during the biological night when the circadian system is promoting sleep adversely influences the success of weight loss therapy. In contrast, restricting EI to a short window during waking hours and extending the length of the overnight fast (i.e., time restricted feeding, TRF) may be a practical and useful strategy for promoting weight loss and weight maintenance. However, potential benefits of adding TRF to a weight loss program have yet to be evaluated in a well-controlled clinical study. The overall objective of this proposal is to provide a foundation to inform the design of a future large-scale trial to evaluate the efficacy of TRF in generating weight loss. The investigators overall hypothesis is that feasibility, adherence, and acceptability of a weight loss intervention using TRF in the setting of a reduced calorie diet (RCD) - RCD+TRF - will be similar to compliance with an intervention using a reduced calorie diet alone (RCD), suggesting acceptability for a future large-scale trial. In this 12-week pilot and feasibility study, 30 overweight and obese individuals will be randomized 1:1 to RCD+TRF (EI restricted to a 10-hour window starting 1 hour from habitual waking time) or standard RCD (no restriction on feeding duration). Additional follow-up will occur at 6 months to collect pilot data on weight maintenance. Measures include feasibility, acceptability and adherence to the interventions, body weight, body composition (Dual-energy X-ray absorptiometry (DXA)), EI (smart phone application), physical activity (PA, accelerometery), glucose variability (continuous glucose monitoring, CGM), sleep (questionnaires and polysomnography), and nocturnal substrate metabolism (room calorimetry). The specific aims (SA) are as follows:

Specific Aim 1a. To evaluate the feasibility and acceptability of a 12-week TRF intervention compared to a standard dietary weight loss intervention (i.e. RCD). Feasibility of enrollment and retention, and acceptability of the intervention will be assessed in adults with obesity meeting inclusion/exclusion criteria proposed for the future large-scale trial. The investigators will assess adherence to the weight loss programs, as measured objectively with a novel smartphone application and verified with CGM data, and subjectively with the use of questionnaires.

Specific Aim 1b. To assess the efficacy of RCD+TRF compared to RCD alone in producing weight loss at 12 weeks and reducing the risk of weight regain after 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females with a BMI of 27-45 kg/m2 and weight stable over the previous 6 months;
* Age, 18-50 years old;
* Passing medical and physical screening, and analysis of blood and urine screening samples;
* Typical eating duration >12 hours per day (assessed by questionnaires);
* Own a smartphone

Exclusion Criteria:

* Pregnancy or lactation for women (women who are >6 months postpartum with no plans of becoming pregnant in the next year and who are not currently lactating can be included; oral contraceptives will be allowed if medication has been consistent for the prior 6 months)
* Postmenopausal women (menopausal status will be assessed during the history and physical, with requirement of self-reported regular menstrual cycles for the last year; women who have undergone hysterectomy but with ovaries in place who continue to have regular menstrual symptoms can be included)
* Being considered unsafe to participate as determined by the study physician;
* History of cardiovascular disease, diabetes, uncontrolled hypertension, untreated thyroid, renal, hepatic diseases, dyslipidemia or any other medical condition affecting weight or lipid metabolism;
* History of human immunodeficiency virus or hepatitis B or C (self-report);
* Taking medications affecting weight or energy intake/energy expenditure in the last 6 months, including weight loss medications, antipsychotic drugs or other medications as determined by the study physician;
* Having abnormal blood chemistry (eGFR<45mL/min, AST or ALT >3 times the upper limit of normal) or as deemed significant by the study physician;
* Being a smoker or having been a smoker in the 3 months prior to their screening visit;
* Working night shifts;
* Extreme early or extreme late chronotype as determined by the Munich Chronotype questionnaire37;
* Night eating syndrome (at least 25% of food intake is consumed after the evening meal and/or at least two episodes of nocturnal eating per week) as assessed with meal pattern assessment questionnaire;
* For participants completing the PSG studies, greater than moderate sleep apnea (score high risk ≥ 2 or more categories on the Berlin Questionnaire). Participants completing the primary weight loss intervention will not be excluded based on Berlin OSA risk scores.
* For participants completing the PSG studies, use of medications affecting sleep (benzodiazepines and other sleep aids, as determined by study physician). Participants completing the primary weight loss intervention will not be excluded based on use of medications affecting sleep.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Thomas, MD, Principal Investigator — University of Colorado Anschutz Health and Wellness Center
Locations (1):
- University of Colorado Anschutz Health and Wellness Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas EA, Zaman A, Sloggett KJ, Steinke S, Grau L, Catenacci VA, Cornier MA, Rynders CA. Early time-restricted eating compared with daily caloric restriction: A randomized trial in adults with obesity. Obesity (Silver Spring). 2022 May;30(5):1027-1038. doi: 10.1002/oby.23420. PMID 35470974
- [Derived] Zaman A, Sloggett KJ, Caldwell AE, Catenacci VA, Cornier MA, Grau L, Vetter C, Rynders CA, Thomas EA. The effects of the COVID-19 pandemic on weight loss in participants in a behavioral weight-loss intervention. Obesity (Silver Spring). 2022 May;30(5):1015-1026. doi: 10.1002/oby.23399. Epub 2022 Apr 12. PMID 35118814

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reduced Calorie Diet (RCD) | Time Restricted Feeding (TRF)
Started | 40 | 41
Completed | 31 | 32
Not Completed | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reduced Calorie Diet (RCD) | Time Restricted Feeding (TRF) | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 41 | 81
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (7.8) | 38.3 (7.9) | 38 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 69
  Male | 5 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 32 | 35 | 67
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 30 | 36 | 66
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 40 | 41 | 81

OUTCOME MEASURES:

1. Primary Outcome: Changes in Body Weight
Description: Body weight will be measured via clinic scale.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Reduced Calorie Diet (RCD) | Time Restricted Feeding (TRF)
Number analyzed (Participants) | 27 | 33
kg | -5.1 (3.2) | -6.2 (4.1)

2. Secondary Outcome: Changes in Fat Mass
Description: Body composition will be assessed with dual-energy x-ray absorptiometry (DXA).
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Reduced Calorie Diet (RCD) | Time Restricted Feeding (TRF)
Number analyzed (Participants) | 23 | 24
kg | -2.1 (2.6) | -2.8 (1.8)

3. Secondary Outcome: Changes in Objectively Measured Energy Intake (Camera)
Description: All energy intake events will be recorded using the camera function on a cell phone application
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Reduced Calorie Diet (RCD) | Time Restricted Feeding (TRF)
Number analyzed (Participants) | 32 | 32
kcal | -612.2 (476) | -647.3 (773)

4. Secondary Outcome: Changes in Physical Activity
Description: Step count will be measured with activity monitors.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | Reduced Calorie Diet (RCD) | Time Restricted Feeding (TRF)
Number analyzed (Participants) | 34 | 35
steps/day | 576 (3172) | 596 (2731)

5. Secondary Outcome: Changes in Sedentary Behavior
Description: Sitting time will be measured with activity monitors.
Time Frame: Baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Reduced Calorie Diet (RCD) | Time Restricted Feeding (TRF)
Number analyzed (Participants) | 34 | 35
minutes/day | -19.8 (88) | -0.77 (82)

6. Other Pre Specified Outcome: 6 Month Post-Intervention Follow-Up Body Weight
Description: Body weight will be measured via clinic scale at 6 months post-intervention
Time Frame: 24 weeks after completion of the 12-week intervention (i.e. at week 36)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Reduced Calorie Diet (RCD) | Time Restricted Feeding (TRF)
Number analyzed (Participants) | 30 | 30
kg | -4.3 (5.3) | -4.9 (5.3)

7. Other Pre Specified Outcome: 6 Month Post-Intervention Follow-Up Fat Mass
Description: Body composition will be assessed with dual-energy x-ray absorptiometry (DXA).
Time Frame: 24 weeks after completion of the 12-week intervention (i.e. at week 36)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Reduced Calorie Diet (RCD) | Time Restricted Feeding (TRF)
Number analyzed (Participants) | 30 | 30
kg | -2.6 (4.4) | -3.5 (4)

ADVERSE EVENTS:
Time Frame: 39 weeks
Arm/Group | Reduced Calorie Diet (RCD) | Time Restricted Feeding (TRF)
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/41
Other Adverse Events (participants affected / at risk) | 0/40 | 0/41

LIMITATIONS AND CAVEATS:
This study was interrupted by the COVID-19 pandemic and the originally planned method for obtaining body weight at 12 weeks (DXA) could not be performed in the 3rd cohort of participants, so home scale weights were used instead.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT03571048/Prot_SAP_000.pdf